CLINICAL TRIAL: NCT05035017
Title: Clinical Validation of the Apollo Daily Disposable Soft Contact Lenses
Status: Completed | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-20-63
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2022-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (2):
- Test Lens, then Control Lens (Experimental): Participants wore Test Lens for 2 days, and then Control Lens for 2 days
  Interventions: Device: Test Lens; Device: Control Lens
- Control Lens, then Test Lens (Active Comparator): Participants wore Control Lens for 2 days, and then Test Lens for 2 days
  Interventions: Device: Test Lens; Device: Control Lens

INTERVENTIONS:
Device: Test Lens — Daily disposable with modified lens design for 2 days
Device: Control Lens — Daily disposable lens for 2 days

SUMMARY:
The purpose of this study was to confirm the design specifications of a Test lens and validate its clinical performance.

DETAILED DESCRIPTION:
This was a double-masked, randomized, bilateral two-day crossover, dispensing study design. Subjects were randomized to wear the Test lens or Control lens bilaterally in random order and on a daily wear, single-use basis for a period of 2 days each.

ELIGIBILITY:
Inclusion Criteria:

* Has had a self-reported oculo-visual examination in the last two years.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is an adapted soft contact lens wearer, having worn contact lenses for a minimum 4 weeks prior to the study
* Has spectacle cylinder ≤1.00D in both eyes.
* Has spherical contact lens power requirement between -1.00D and -6.00D in both eyes.
* Has manifest refraction visual acuities (VA) equal to or better than logMAR equivalent of 20/20 in each eye.
* Wears CLs in both eyes (monovision acceptable, but not monofit)
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination
* Is willing to wear the study contact lenses for a minimum 8 hours on at least two consecutive days for each study pair.

Exclusion Criteria:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any concomitant systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye-related clinical or research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Optometry, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Lens, Then Control Lens: Participants wore Test Lens for 2 days (Period 1), and then Control Lens for 2 days (Period 2)
- Control Lens, Then Test Lens: Participants wore Control Lens for 2 days (Period 1), and then Test Lens for 2 days (Period 2)
Period: Period 1 (2 Days)
Arm/Group | Test Lens, Then Control Lens | Control Lens, Then Test Lens
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0
Period: Period 2 (2 Days)
Arm/Group | Test Lens, Then Control Lens | Control Lens, Then Test Lens
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All participants who were dispensed lenses and successfully completed the study
Arm/Group | Overall Study
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort With Lens
Description: Participants rated their overall comfort once after 2 days of wear a 0-100 integer scale, where 0=Cannot be tolerated and 100=Excellent comfort.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Test Lens: Participants that received Test lens during either the first or second period of the study.
- Control Lens: Participants that received Control lens during either the first or second period of the study.
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 35 | 35
score on a scale | 86 (15) | 72 (26)

2. Secondary Outcome: Overall Vision Quality
Description: Participant response measured once after 2 days of wear on a 0-100 integer scale, where 0= Unacceptable, 100=Excellent Vision.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 35 | 35
score on a scale | 90 (11) | 91 (11)

3. Secondary Outcome: Overall Lens Fit Acceptance
Description: Measured once after 2 days of wear by investigator on lens fit alone (excludes comfort, vision, orientation) on a 0-4 scale, 0.25 steps, where 0=Can't be worn and 4=Optimum
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 35 | 35
score on a scale | 3.11 (0.66) | 3.09 (0.70)

4. Secondary Outcome: Overall Lens Handling
Description: Participant response on overall handling (insertion, removal, and holding) of contact lenses assessed once after 2 days of wear, on the third day. Measured on a 0-100 integer scale, where 0=Cannot be managed, 100=Excellent handling.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 35 | 35
score on a scale | 88 (15) | 87 (14)

5. Secondary Outcome: Anterior Ocular Health - Corneal Staining Extent
Description: Assessed once after 2 days of wear with slit lamp biomicroscopy and graded on a 0-4 integer scale, where 0=No Staining and 4=>45% of area. Lower values represented a better outcome, e.g., a grading value of 1 would represent less corneal staining than a grade of 4. Locations (central, nasal, temporal, superior, inferior) were graded separately.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Lens | Control Lens
Number analyzed (Participants) | 35 | 35
score on a scale
  Central | 0.10 (0.30) | 0.16 (0.44)
  Nasal | 0.11 (0.32) | 0.14 (0.39)
  Temporal | 0.10 (0.30) | 0.13 (0.34)
  Superior | 0.04 (0.20) | 0.06 (0.23)
  Inferior | 0.39 (0.52) | 0.41 (0.55)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 4 days
Arm/Group | Test Lens | Control Lens
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT05035017/Prot_SAP_000.pdf